CLINICAL TRIAL: NCT06891638
Title: Enhancing Reading Recovery in Aphasia With tDCS and PMT
Brief Title: Enhancing Reading Recovery in Aphasia With tDCS and Phonomotor Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Olga Boukrina, Assistant Director, Center for Stroke Rehabilitation Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-1290-25
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Aphasia
Keywords: Aphasia; Post-stroke rehabilitation; Reading impairment; Language therapy; Transcranial Direct Current Stimulation (tDCS); Phonomotor Treatment (PMT); Brain stimulation therapy; Neurorehabilitation; Randomized controlled trial (RCT); Non-invasive brain stimulation; Neuromodulation; Speech and language therapy
MeSH Terms: conditions — Stroke; Aphasia; Dyslexia; Communication Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early tDCS (Experimental): This group will undergo Active tDCS + PMT for weeks 1-3 and Sham tDCS + PMT for weeks 4-6.
  Interventions: Device: Schedule of tDCS administration
- Late tDCS (Sham Comparator): This group will undergo Sham tDCS + PMT for weeks 1-3 and Active tDCS + PMT for weeks 4-6.
  Interventions: Device: Schedule of tDCS administration
- Interleaved tDCS (Active Comparator): This group will receive PMT + Active/Sham tDCS on alternate days for 6 weeks.
  Interventions: Device: Schedule of tDCS administration

INTERVENTIONS:
Device: Schedule of tDCS administration — This study evaluates the combined effects of Phono-Motor Treatment (PMT) and transcranial direct current stimulation (tDCS) for reading rehabilitation in post-stroke aphasia. Unlike standard speech therapy, this intervention integrates non-invasive brain stimulation to enhance language recovery by modulating neural activity in perilesional areas. We hypothesize that active tDCS will enhance PMT efficacy, leading to greater improvements in reading competence and phonological processing compared to sham tDCS. Through systematic testing across the 3 study arms, we expect to identify the most effective stimulation timing.

SUMMARY:
This study is designed for individuals with aphasia, a language disorder that affects many stroke survivors, making it difficult to read, speak, and understand language. Up to 70% of people with aphasia struggle with reading, which impacts their ability to communicate, work, and engage in daily life.

The study aims to test a new approach to reading rehabilitation by combining Phono-Motor Treatment (PMT), a language therapy adapted to improve reading, with transcranial direct current stimulation (tDCS), a safe and painless brain stimulation technique. tDCS delivers a mild electrical current to the brain, which may enhance learning. This study will assess whether adding tDCS to PMT improves reading therapy outcomes.

DETAILED DESCRIPTION:
This study aims to improve reading rehabilitation for individuals with aphasia, a language disorder that affects many stroke survivors. The goal is to determine whether adding transcranial direct current stimulation (tDCS), a safe and painless brain stimulation technique, to Phono-Motor Treatment (PMT), a language therapy adapted for reading, enhances treatment effectiveness.

Participants will be randomly assigned to one of three treatment groups, each receiving different combinations of PMT and tDCS over six weeks. Some will receive active tDCS at different points in therapy, while others will receive a placebo (sham) version. By comparing how the timing of tDCS affects reading improvement, this study aims to optimize treatment strategies for individuals with aphasia.

Reading and language skills will be assessed before, during, and after treatment using standardized tests to measure progress. The study will take place at two sites: Kessler Foundation and the Medical College of Wisconsin (MCW), where participants will complete therapy sessions.

Findings from this research may help develop more effective and accessible treatments for stroke survivors with aphasia, improving their ability to read and communicate.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (>6 months) left-hemisphere stroke
* Aphasia diagnosis.
* Deficits in reading aloud.

Exclusion Criteria:

* Eye condition not correctable with lenses and interfering with reading (e.g., blindness)
* Severe apraxia of speech or cognitive deficits preventing participation.
* Participation in one-on-one aphasia rehabilitation during the study period.
* Brain disorders other than stroke (such as Alzheimer's Disease or Dementia, Parkinson's Disease, etc)
* Contraindications of tDCS or MRI

  * Skin condition affecting the scull (e.g., psoriasis) or open wounds at the stimulation site.
  * Presence of metallic implants (e.g., cardiac stimulators or pacemakers, cochlear implants)
  * History of ongoing/unmanaged seizers
  * Pregnancy
  * Claustrophobia
  * Inability to lie flat on the back

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Reading aloud accuracy | before treatment, midway through treatment, and immediately after treatment
  Participants will read words and pronounceable pseudowords that appear one at a time on the computer screen. Each testing session will be audio recorded and independently scored by 2 raters, with ties resolved by a 3rd rater.

SECONDARY OUTCOMES:
Reading Comprehension Battery for Aphasia 2nd Edition | before treatment, midway through treatment, and immediately after treatment
  Participants will complete a standardized language assessment.
Western Aphasia Battery | before treatment, midway through treatment, and immediately after treatment
  Participants will complete a standardized language assessment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kessler Foundation, West Orange, New Jersey
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided